CLINICAL TRIAL: NCT03383055
Title: CMV-MVA Triplex Vaccine to Enhance Adaptive NK Cell Reconstitution After Autologous Hematopoietic Cell Transplantation in Patients With Lymphoid Malignancies
Brief Title: CMV-MVA Triplex Vac.Enhance Adap. NK Cell Recon. After Auto HSCT in pt Lymphoid Malig
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017LS091; MT2017-29 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2017-12-11; First posted 2017-12-26 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMV positive cohort (Experimental): CMV-MVA Triplex vaccine administered on days 28 and 56 post-HCT
  Interventions: Biological: CMV-MVA Triplex Vaccine
- CMV negative cohort (Experimental): CMV-MVA Triplex vaccine administered on days 28 and 56 post-HCT
  Interventions: Biological: CMV-MVA Triplex Vaccine

INTERVENTIONS:
Biological: CMV-MVA Triplex Vaccine — * CMV-MVA Triplex vaccine administered on days 28 and 56 post-HCT
  * TDap administered on Day 56

SUMMARY:
This is a prospective, interventional study administering 2 doses of the experimental vaccine (CMV-MVA Triplex) to 20 evaluable patients (10 CMV-seropositive and 10 seronegative) undergoing autologous hematopoietic cell transplantation (HCT) for lymphoma or myeloma on days 28 and 56 post-HCT. The absolute number of adaptive NK cells (CD56dimCD57+NKG2C+) at various days will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Lymphoma or multiple myeloma
* Planned co-enrollment on current (at the time of this study version) or future (opening subsequent to this study) standard of care autologous stem cell transplant protocol.

  * Must meet all eligibility requirements of the co-enrolled parent study
* Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control until at least day 100 post-HCT
* Voluntary written consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* CMV immunoglobulin, valganciclovir, ganciclovir, foscarnet, or other anti-CMV therapy within 3 months before the first vaccine is planned. Acyclovir and valacyclovir are allowed.
* Pregnant or breast feeding. The FDA has not classified this agent into a specified pregnancy category. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
* Planned immunotherapy post-HCT. Proteasome inhibitors and/or immunomodulators, such as but not limited to Lenalidomide or Pomalidomide, used for myeloma maintenance are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Change in the absolute number of CMV-induced adaptive NK cells (CD56dimCD57+NKG2C+) between days 28 and 100 post-auto-HCT in patients with lymphoid malignancies. | Day 28 and Day 100
  Change in the absolute number of CMV-induced adaptive NK cells (CD56dimCD57+NKG2C+) on day 28 (pre first vaccine) and day 100 (~1 month after second vaccine) post-auto- HCT in patients with lymphoid malignancies.

SECONDARY OUTCOMES:
Change in absolute Number of CMV-induced adaptive NK Cells | Day 28 and Day 100
  Change in absolute number of total NK and NK/T cells between days 28 (first vaccine) and day 100 (~1 month after second vaccine) post-auto-HCT in patients with lymphoid malignancies (lymphoma and myeloma).
Response to CMV-MVA Triplex vaccine in CMV seropositive vs. seronegative patients | Day 28 and Day 100
  Change in the absolute number of adaptive NK cells between day 28 post-transplant and day 100.
Progression Free Survival (PFS) | 1 Year
  Incidence of progression-free survival at 1 year in patients receiving CMV-MVA Triplex vaccine with historical controls
Response to CMV-MVA Triplex vaccine in lymphoma vs. myeloma patients | Day 28 and Day 100
  Change in the absolute number of adaptive NK cells between day 28 post-transplant and day 100.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Rashidi, MD, PhD, Principal Investigator — University of Minnesota Hematology, Oncology and Transplantation Department of Medicine
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03383055/ICF_000.pdf